CLINICAL TRIAL: NCT00576121
Title: Measurement of Matrix Metalloproteinase Activation Post Myocardial Infarction
Status: Withdrawn | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0610001945
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Left ventricular ejection fraction (LVEF) patients will be compared at two time-points, 2-5 days and 4 weeks after acute MI.
- 2: End-diastolic volume (LVEDV) patients will be compared at two time-points, 2-5 days and 4 weeks after acute MI.
- 3: End-systolic volume (LVESV) patients will be compared at two time-points, 2-5 days and 4 weeks after acute MI.

SUMMARY:
This study is designed to look at the measurement and prediction of changes in the heart following a heart attack.

DETAILED DESCRIPTION:
Patients who are admitted to Yale New Haven Hospital with first acute myocardial infarction within the onset of 12 hours of symptoms will be eligible for this study and referred by their physician for this study. Subjects will be screened with medical interview and physical exam for eligibility. Clinical data will be obtained for demographic purposes including: EKG upon admission, serum cardiac markers, basic metabolic panel, cardiac catheterization report and recent echocardiography report. All standard medications will be allowed which include diuretics, ACE/Ang-II inhibitors, nitrates/hydralazine, digoxin, low dose aspirin, beta-blockers, calcium channel antagonists, anticoagulants and anti-arrhythmic agents.

A 10cc blood sample will be drawn from a peripheral vein at 3 days post myocardial infarction into chilled EDTA tubes, plasma decanted and placed at -70 degrees C until MMP/TIMP assays are performed. These samples will be sent to collaborators at the Medical University of South Carolina for high sensitivity plasma assays developed at MUSC for MMP-1, -13, -8, -2, -9 and TIMP-1, -2, -4. [1] These assays will be performed in Core C and detailed description of specificity of these measurements is described. In addition, indices of collagen synthesis and degradation, through the use of telopeptide measurements will be measured in these plasma samples.

Nitroglycerin resting Tl-201 myocardial perfusion imaging will be performed between 2-5 days after myocardial infarction. Subjects will have a peripheral intravenous line placed and will be injected with 2.5-3.5mCi of Tl-201. The Tl-201 given will be a slightly lower dosage than the standard clinical protocol of Yale New Haven Hospital nuclear cardiology lab because of improved reconstruction algorithms with CT will allow lower doses of radioactive isotopes. Resting myocardial perfusion images will be acquired 5 minutes post-injection on a multislice helical SPECT/CT (GE Infinia Hawkeye) followed by a CT scan. A redistribution image will be performed 4 hours after thallium administration. Each SPECT scan will take approximately 25 minutes. Perfusion defect size will be quantified using the Yale C-Q method previously described [2].

Transthoracic echocardiography will be performed at 2-5 days post-MI and 28 days after MI in standard apical and parasternal views using a commercial ultrasound system either Phillips 7500 or IE33 ultrasound imaging system with an S3 transducer. The transducer will be placed on the apical and/or parasternal location on the chest and ECG-gated images will be obtained during a breath hold. Each acquisition will be performed in zoom mode at 40 Hz, over the entire LV in 4 cardiac cycles with 40 frames per cardiac cycle. Image data will be captured in digital form and will be backed up on DVDs. NOTE: No patient HIPPA data will be saved on the DVD. Left ventricular ejection fraction (LVEF), end-diastolic volume (LVEDV), and end-systolic volume (LVESV) will be measured. The echocardiograms will be used to determine LV mass, LV cavity size and regional thickening. Patients will undergo MRI with gadolinium contrast in the GE Signa 1.5 tesla magnetic resonance image scanner located in the Yale-New Haven Hospital MRI Center, using standard ECG-gated cine gradient echo, and echo-planar, phase contrast and MR tagged imaging sequences.

Electrocardiographic monitoring will be maintained during the magnetic resonance imaging. MRI scans will occur between 2-5 days post-MI.

The first acquisitions to be performed will be combined cine-gradient echo/cine phase velocity approach that will obtain both the magnitude images required for our segmentation and shape-based tracking as well as contrast data for finding midwall myocardial velocities in a single image acquisition. This sequence will yield adjacent 5 mm thick axial images with in plane resolution of approximately 1.6mm x 1.6mm. We will acquire 16-20 cardiac phase per location. Patients will receive 0.1 mmol/kg of standard gadolinium contrast in a peripheral IV. The acquisition will apply inversion recovery preparatory pulse to null normal myocardium, followed by a segmented k-space gradient echo acquisition. We anticipate that all of the proposed magnetic resonance imaging for each subject will be completed within 2 hours. The technologist or doctor operating the scanner will be able to see the subject. The operator will maintain contact by voice with the subjects.

None of the aforementioned procedures are considered experimental and individually, may or may not be part of the subjects' standard of care post myocardial infarction. During each part of the step of image acquisition, there will be a physician present. All data will be transferred via network to the image processing laboratory for analysis and will not include any projected personal information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myocardial infarction characterized by (1) greater than 30 minutes of chest pain; (2) ST elevation in 2 contiguous leads greater than 2mV; and (3) elevated serum markers greater than three times the normal value.
* Males or females 18 years of age or older.
* Adequate intravenous access in one arm.
* Willing to comply with the requirements of the protocol.
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* History of significant co-morbidity requiring hospitalization separate from acute myocardial infarction (i.e. metastatic cancer).
* History of/current structural heart disease.
* Arrhythmia
* History of previous myocardial infarction
* History of coronary revascularization
* Cardiogenic shock
* Hypotension
* Renal failure (creatinine >2mg/dl) or hyperkalemia (serum potassium > 5.5mg/dl)
* History of allergic reaction to gadolinium
* Contraindication to undergo MR imaging (pacemaker, metallic implants, etc)
* History of claustrophobia
* Pregnant or breast-feeding, or (if pre-menopausal), not practicing acceptable method of birth control.
* History of any other conditions, which in the judgment of the investigator, are likely to hinder or confuse study conduct or to pose a safety concern to the patient.
* Resting HR >110
* Chronic tetracycline or doxycycline use
* Ongoing/active rheumatic disease requiring significant anti-inflammatory agents, steroids or immunosuppression
* Not capable of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by a physician referral into the study. Patients will be referred to the study by the cardiologist in the cardiac catheterization lab at Yale New Haven Hospital. Patient recruitment will be limited to patients who are English speakers. Informed consent will be obtained by Dr. Albert Sinusas, MD.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To predict left ventricular remodeling after myocardial infarction using serum matrix metalloproteinase measurement with Tl201 SPECT/CT hybrid imaging and MRI. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Sinusas, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] Lindsey ML. MMP induction and inhibition in myocardial infarction. Heart Fail Rev. 2004 Jan;9(1):7-19. doi: 10.1023/B:HREV.0000011390.44039.b7. PMID 14739764
- [Background] Cohn JN, Ferrari R, Sharpe N. Cardiac remodeling--concepts and clinical implications: a consensus paper from an international forum on cardiac remodeling. Behalf of an International Forum on Cardiac Remodeling. J Am Coll Cardiol. 2000 Mar 1;35(3):569-82. doi: 10.1016/s0735-1097(99)00630-0. PMID 10716457
- [Background] Wilson EM, Moainie SL, Baskin JM, Lowry AS, Deschamps AM, Mukherjee R, Guy TS, St John-Sutton MG, Gorman JH 3rd, Edmunds LH Jr, Gorman RC, Spinale FG. Region- and type-specific induction of matrix metalloproteinases in post-myocardial infarction remodeling. Circulation. 2003 Jun 10;107(22):2857-63. doi: 10.1161/01.CIR.0000068375.40887.FA. Epub 2003 May 27. PMID 12771000
- [Background] Kai H, Ikeda H, Yasukawa H, Kai M, Seki Y, Kuwahara F, Ueno T, Sugi K, Imaizumi T. Peripheral blood levels of matrix metalloproteases-2 and -9 are elevated in patients with acute coronary syndromes. J Am Coll Cardiol. 1998 Aug;32(2):368-72. doi: 10.1016/s0735-1097(98)00250-2. PMID 9708462
- [Background] Bradham WS, Gunasinghe H, Holder JR, Multani M, Killip D, Anderson M, Meyer D, Spencer WH 3rd, Torre-Amione G, Spinale FG. Release of matrix metalloproteinases following alcohol septal ablation in hypertrophic obstructive cardiomyopathy. J Am Coll Cardiol. 2002 Dec 18;40(12):2165-73. doi: 10.1016/s0735-1097(02)02595-0. PMID 12505230
- [Background] Spinale FG. Matrix metalloproteinases: regulation and dysregulation in the failing heart. Circ Res. 2002 Mar 22;90(5):520-30. doi: 10.1161/01.res.0000013290.12884.a3. PMID 11909815
- [Background] Mukherjee R, Brinsa TA, Dowdy KB, Scott AA, Baskin JM, Deschamps AM, Lowry AS, Escobar GP, Lucas DG, Yarbrough WM, Zile MR, Spinale FG. Myocardial infarct expansion and matrix metalloproteinase inhibition. Circulation. 2003 Feb 4;107(4):618-25. doi: 10.1161/01.cir.0000046449.36178.00. PMID 12566376
- [Background] Ducharme A, Frantz S, Aikawa M, Rabkin E, Lindsey M, Rohde LE, Schoen FJ, Kelly RA, Werb Z, Libby P, Lee RT. Targeted deletion of matrix metalloproteinase-9 attenuates left ventricular enlargement and collagen accumulation after experimental myocardial infarction. J Clin Invest. 2000 Jul;106(1):55-62. doi: 10.1172/JCI8768. PMID 10880048
- [Background] Creemers EE, Davis JN, Parkhurst AM, Leenders P, Dowdy KB, Hapke E, Hauet AM, Escobar PG, Cleutjens JP, Smits JF, Daemen MJ, Zile MR, Spinale FG. Deficiency of TIMP-1 exacerbates LV remodeling after myocardial infarction in mice. Am J Physiol Heart Circ Physiol. 2003 Jan;284(1):H364-71. doi: 10.1152/ajpheart.00511.2002. Epub 2002 Sep 26. PMID 12388239
- [Background] Lindsey ML, Escobar GP, Dobrucki LW, Goshorn DK, Bouges S, Mingoia JT, McClister DM Jr, Su H, Gannon J, MacGillivray C, Lee RT, Sinusas AJ, Spinale FG. Matrix metalloproteinase-9 gene deletion facilitates angiogenesis after myocardial infarction. Am J Physiol Heart Circ Physiol. 2006 Jan;290(1):H232-9. doi: 10.1152/ajpheart.00457.2005. Epub 2005 Aug 26. PMID 16126817
- [Background] Su H, Spinale FG, Dobrucki LW, Song J, Hua J, Sweterlitsch S, Dione DP, Cavaliere P, Chow C, Bourke BN, Hu XY, Azure M, Yalamanchili P, Liu R, Cheesman EH, Robinson S, Edwards DS, Sinusas AJ. Noninvasive targeted imaging of matrix metalloproteinase activation in a murine model of postinfarction remodeling. Circulation. 2005 Nov 15;112(20):3157-67. doi: 10.1161/CIRCULATIONAHA.105.583021. Epub 2005 Nov 7. PMID 16275862
- [Background] Higo S, Uematsu M, Yamagishi M, Ishibashi-Ueda H, Awata M, Morozumi T, Ohara T, Nanto S, Nagata S. Elevation of plasma matrix metalloproteinase-9 in the culprit coronary artery in patients with acute myocardial infarction: clinical evidence from distal protection. Circ J. 2005 Oct;69(10):1180-5. doi: 10.1253/circj.69.1180. PMID 16195613
- [Background] Hojo Y, Ikeda U, Katsuki Ta, Mizuno O, Fujikawa H, Shimada K. Matrix metalloproteinase expression in the coronary circulation induced by coronary angioplasty. Atherosclerosis. 2002 Mar;161(1):185-92. doi: 10.1016/s0021-9150(01)00615-3. PMID 11882331
- [Background] Hojo Y, Ikeda U, Ueno S, Arakawa H, Shimada K. Expression of matrix metalloproteinases in patients with acute myocardial infarction. Jpn Circ J. 2001 Feb;65(2):71-5. doi: 10.1253/jcj.65.71. PMID 11216828
- [Background] Sundstrom J, Evans JC, Benjamin EJ, Levy D, Larson MG, Sawyer DB, Siwik DA, Colucci WS, Sutherland P, Wilson PW, Vasan RS. Relations of plasma matrix metalloproteinase-9 to clinical cardiovascular risk factors and echocardiographic left ventricular measures: the Framingham Heart Study. Circulation. 2004 Jun 15;109(23):2850-6. doi: 10.1161/01.CIR.0000129318.79570.84. Epub 2004 Jun 1. PMID 15173025
- [Background] Sundstrom J, Evans JC, Benjamin EJ, Levy D, Larson MG, Sawyer DB, Siwik DA, Colucci WS, Wilson PW, Vasan RS. Relations of plasma total TIMP-1 levels to cardiovascular risk factors and echocardiographic measures: the Framingham heart study. Eur Heart J. 2004 Sep;25(17):1509-16. doi: 10.1016/j.ehj.2004.05.029. PMID 15342170
- [Background] Kaden JJ, Dempfle CE, Sueselbeck T, Brueckmann M, Poerner TC, Haghi D, Haase KK, Borggrefe M. Time-dependent changes in the plasma concentration of matrix metalloproteinase 9 after acute myocardial infarction. Cardiology. 2003;99(3):140-4. doi: 10.1159/000070670. PMID 12824721
- [Background] Webb CS, Bonnema DD, Ahmed SH, Leonardi AH, McClure CD, Clark LL, Stroud RE, Corn WC, Finklea L, Zile MR, Spinale FG. Specific temporal profile of matrix metalloproteinase release occurs in patients after myocardial infarction: relation to left ventricular remodeling. Circulation. 2006 Sep 5;114(10):1020-7. doi: 10.1161/CIRCULATIONAHA.105.600353. Epub 2006 Aug 21. PMID 16923753
- [Background] Choi JY, Moon DH, Lee CW, Shin JW, Park SW, Hong MK, Song JK, Park SJ, Lee HK. Prediction of left ventricular dilatation with thallium-201 SPET imaging after primary angioplasty in patients with acute myocardial infarction. Eur J Nucl Med Mol Imaging. 2002 Jun;29(6):728-34. doi: 10.1007/s00259-002-0800-y. Epub 2002 Apr 6. PMID 12029545
- [Background] Oudiz RJ, Smith DE, Pollak AJ, Mena I, Shapiro SM, Ginzton LE, Narahara KA. Nitrate-enhanced thallium 201 single-photon emission computed tomography imaging in hibernating myocardium. Am Heart J. 1999 Aug;138(2 Pt 1):369-75. doi: 10.1016/s0002-8703(99)70127-4. PMID 10426854
- [Background] Watzinger N, Lund GK, Higgins CB, Wendland MF, Weinmann HJ, Saeed M. The potential of contrast-enhanced magnetic resonance imaging for predicting left ventricular remodeling. J Magn Reson Imaging. 2002 Dec;16(6):633-40. doi: 10.1002/jmri.10206. PMID 12451576
- [Background] Schroeder AP, Houlind K, Pedersen EM, Nielsen TT, Egeblad H. Serial magnetic resonance imaging of global and regional left ventricular remodeling during 1 year after acute myocardial infarction. Cardiology. 2001;96(2):106-14. doi: 10.1159/000049092. PMID 11740140
- [Background] Wellnhofer E, Olariu A, Klein C, Grafe M, Wahl A, Fleck E, Nagel E. Magnetic resonance low-dose dobutamine test is superior to SCAR quantification for the prediction of functional recovery. Circulation. 2004 May 11;109(18):2172-4. doi: 10.1161/01.CIR.0000128862.34201.74. Epub 2004 Apr 26. PMID 15117834
- [Background] Hombach V, Grebe O, Merkle N, Waldenmaier S, Hoher M, Kochs M, Wohrle J, Kestler HA. Sequelae of acute myocardial infarction regarding cardiac structure and function and their prognostic significance as assessed by magnetic resonance imaging. Eur Heart J. 2005 Mar;26(6):549-57. doi: 10.1093/eurheartj/ehi147. Epub 2005 Feb 15. PMID 15713695
- [Background] Bucciarelli-Ducci C, Wu E, Lee DC, Holly TA, Klocke FJ, Bonow RO. Contrast-enhanced cardiac magnetic resonance in the evaluation of myocardial infarction and myocardial viability in patients with ischemic heart disease. Curr Probl Cardiol. 2006 Feb;31(2):128-68. doi: 10.1016/j.cpcardiol.2005.10.002. No abstract available. PMID 16413381
- [Background] Soejima H, Ogawa H, Sakamoto T, Miyamoto S, Kajiwara I, Kojima S, Hokamaki J, Sugiyama S, Yoshimura M, Suefuji H, Miyao Y, Fujimoto K, Miyagi H, Kishikawa H. Increased serum matrix metalloproteinase-1 concentration predicts advanced left ventricular remodeling in patients with acute myocardial infarction. Circ J. 2003 Apr;67(4):301-4. doi: 10.1253/circj.67.301. PMID 12655159